CLINICAL TRIAL: NCT06907017
Title: First In Human Clinical Study of the CorWave Left Ventricular Assist System for the Treatment of Patients With Advanced Heart Failure
Brief Title: CorWave LVAS FIH Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CorWave (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-2023-CTN-01360-1
Record Dates: First submitted 2025-03-21; First posted 2025-04-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects implanted with CorWave LVAD (Experimental)
  Interventions: Device: LVAS

INTERVENTIONS:
Device: LVAS — Implantation and use of the CorWave LVAS to evaluate the safety and effectiveness of the CorWave LVAD to treat advanced left ventricular heart failure.

SUMMARY:
The study is a prospective, multi-center, non-randomized trial to evaluate the safety and effectiveness of the CorWave LVAS for the treatment of advanced heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative has signed Informed Consent Form
* Age > 18 and < 75 years old
* Body Surface Area (BSA) ≥ 1.2 m2
* Left Ventricular Ejection Fraction (LVEF) ≤ 35%
* Inotrope dependent OR
* Cardiac Index (CI) < 2.2 L/min/m2, while not on inotropes and subjects must also meet one of the following criteria:

  * On Guideline Directed Medical Therapy (GDMT) for at least 45 out of the last 60 days and are failing to respond.
  * Advanced heart failure (Class III or Class IV for at least 14 days AND support from short term mechanical circulatory support for up to 7 days).
* Females of childbearing age must agree to use adequate contraception.
* Patient must be eligible for heart transplantation.

Exclusion Criteria:

* Heart failure (HF) due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy.
* Technical obstacles which pose an inordinately high surgical risk, in the judgment of the Investigator
* Ongoing mechanical circulatory support (MCS) other than IABP or micro axial pumps
* INTERMACS Class I patients
* Subject is on a ventilator
* Subject is pregnant or breastfeeding
* Presence of a mechanical aortic valve that will not be converted to a bioprosthesis at the time of LVAD implant
* History of any organ transplant
* Platelet count < 100,000/μl
* Psychiatric disease/disorder, illicit drug use, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAD management
* History of confirmed untreated abdominal aortic aneurysm (AAA) > 5 cm in diameter within 6 months of enrollment
* Presence of an active, uncontrolled infection
* Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the patient's health status
* Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:
* An INR ≥ 2.0 not due to anticoagulation therapy
* Total bilirubin > 43 µmol/L (2.5 mg/dL), liver function tests greater than 3 times the establish laboratory normal, including Serum Albumin below 3.5 g/dl, shock liver, or biopsy proven liver cirrhosis
* History of severe chronic obstructive pulmonary disease (COPD) and restrictive disease (fibrosis); FEV1 < 50%, a total FEV1 below 1000 mL and a DLCO < 50% predicted.
* Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
* History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 50%) uncorrected carotid stenosis
* Serum creatinine ≥ 221 µmol/L (2.5 mg/dL) or the need for chronic renal replacement therapy.
* Ongoing patient malnutrition evidenced by nonintentional weight loss of greater than 5% of body mass in the previous 30 days, prealbumin < 16 mg/dL, or Mini Nutritional Assessment score < 17.
* Poorly controlled diabetes mellitus or a hemoglobin A1c > 8.5%.
* Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration.
* Patient has severe aortic insufficiency without plans for correction during pump implant.
* Planned Bi-VAD support prior to enrollment.
* Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia.
* Participation in any other clinical investigation that is likely to confound study results or affect the study.
* Any condition other than HF that could limit survival to less than 12 months.
* Acute myocardial infarction within 14 days of implant as diagnosed by ST elevation (STEMI) changes on ECG, diagnostic biomarkers, and hemodynamic abnormalities. Planned or carried out coronary revascularizations (including PCI requiring (dual) antiplatelet therapies).
* Pulmonary embolus within 6 weeks of implant as documented by computed tomography (CT) scan or nuclear scan.
* Subject is unwilling or unable to comply with trial requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Survival post-implant | 30 days
  Survival at 30 days post index procedure.
Freedom from adverse events associated with CorWave LVAD | 30 days
  Freedom from adverse events associated with the use of the CorWave LVAD through 30 days post LVAD implant defined as non-surgical bleeding, infection, disabling stroke and pump malfunction, as defined by INTERMACS.

SECONDARY OUTCOMES:
Overall survival | up to 2 years
  Survival to transplant or of LVAD support
Freedom from non-surgical bleeding | 180 days
  Freedom from non-surgical bleeding (as defined by INTERMACS)
Freedom from infection | 180 days
  Freedom from infection (as defined by INTERMACS)
Freedom from debilitating stroke | 180 days
  Freedom from debilitating stroke (Modified Rankin Score >3) at 180 days
Health-related Quality of Life | up to 2 years
  Quality of Life measured by EuroQoL (EQ-5D)
Health-related Quality of Life | up to 2 years
  Health-related quaulity of life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Neurocognitive function | up to 2 years
  Neurocognitive function indicated by the Trail-making B test
Functional status | up to 2 years
  Functional status as measured by NYHA classification
Functional status | up to 2 years
  Measured by 6-minute walk test
Adverse Events rates | up to 2 years
  Adverse Events rates, as defined per INTERMACS

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Bayside Health, Melbourne, Victoria